CLINICAL TRIAL: NCT02496897
Title: A Phase I, Randomized, Double-blind, Placebo-controlled, Multi-centre, Ascending-dose Trial to Evaluate the Safety, Tolerability and Immunogenicity of Vaccine FP-02.2 in HBeAg-negative Hepatitis B Patients as an add-on Treatment to Entecavir or Tenofovir.
Brief Title: Phase I Safety and Immunogenicity of FP-02.2 in Chronic Hepatitis B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Altimmune, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FP02.2_CS_01
Record Dates: First submitted 2015-07-06; First posted 2015-07-14 (Estimated); Results first posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- FP-02.2 Low Dose (Experimental): A low dose (150 µg/peptide) of the FP-02.2 vaccine administered by IM injection on Days 1, 29, and 57.
  Interventions: Biological: FP-02.2 Vaccine
- FP-02.2 High Dose (Experimental): A high dose (500 µg/peptide) of the FP-02.2 vaccine administered by IM injection on Days 1, 29, and 57.
  Interventions: Biological: FP-02.2 Vaccine
- FP-02.2 Low Dose with IC31® Adjuvant (Experimental): A low dose (150 µg/peptide) of the FP-02.2 vaccine with IC31® Adjuvant administered by IM injection on Days 1, 29, and 57.
  Interventions: Biological: FP-02.2 Vaccine; Other: IC31® Adjuvant
- FP-02.2 High Dose with IC31® Adjuvant (Experimental): A high dose (500 µg/peptide) of the FP-02.2 vaccine with IC31® Adjuvant administered by IM injection on Days 1, 29, and 57.
  Interventions: Biological: FP-02.2 Vaccine; Other: IC31® Adjuvant
- Placebo (Placebo Comparator): Placebo administered by IM injection on Days 1, 29, and 57.
  Interventions: Other: Placebo
- IC31® Adjuvant (Experimental): IC31® Adjuvant alone administered by IM injection on Days 1, 29, and 57.
  Interventions: Other: IC31® Adjuvant

INTERVENTIONS:
Biological: FP-02.2 Vaccine — Synthetic Peptide Hepatitis B Vaccine
  Arms: FP-02.2 High Dose; FP-02.2 High Dose with IC31® Adjuvant; FP-02.2 Low Dose; FP-02.2 Low Dose with IC31® Adjuvant
Other: Placebo — Placebo
  Arms: Placebo
Other: IC31® Adjuvant — IC31® Adjuvant
  Arms: FP-02.2 High Dose with IC31® Adjuvant; FP-02.2 Low Dose with IC31® Adjuvant; IC31® Adjuvant

SUMMARY:
This study evaluates the safety and immunogenicity of FP-02.2, a new therapeutic Hepatitis B vaccine, administered as an add-on therapy to entecavir or tenofovir.

DETAILED DESCRIPTION:
This study evaluates the safety and immunogenicity of FP-02.2, a new therapeutic Hepatitis B vaccine, administered as an add-on therapy to entecavir or tenofovir. HBeAg-negative subjects will be randomized to receive low or high dose vaccine, in the presence or absence of IC31® adjuvant, or to receive placebo or IC31® adjuvant alone.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18-65 years.
2. Diagnosed with chronic hepatitis B defined as HBsAg positive for at least 24 months.
3. Subject has received entecavir or tenofovir for at least 2 years with a stable dose for at least 6 months prior to screening.
4. HBeAg negative for at least 2 years prior to inclusion in the study.
5. HBV DNA <50 IU/mL for ≥ 12 months
6. ALT/AST ≤ 1.5 x ULN via the local laboratory at the Screening Visit
7. Able to give written informed consent to participate
8. Females should fulfil one of the following criteria:

   1. At least one year menopausal
   2. Surgically sterile
   3. Same-sex relationship
   4. WOCBP not surgically sterilized or with laboratory confirmed menopausal status are required to use a highly effective contraceptive measure with low used dependency from screening until one menstrual cycle after the last dose of IMP (Day 58) such as:

      * Combined (oestrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation
      * Progestogen-only hormonal contraception implants associated with inhibition of ovulation
      * Intrauterine device (IUD)
      * Intrauterine hormone-releasing system (IUS)
      * Bilateral tubal occlusion
      * Vasectomised partner - must have had medical assessment of successful surgery.

From screening until one menstrual cycle after the last dose of IMP (day 57).

Subjects who practice true abstinence or who exclusively have same sex partners need not use contraception, provided it is in line with their preferred and usual lifestyle. Periodic abstinence (eg calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Should any such subject stop practicing true abstinence, they must use contraception as described above.

Males should fulfil one of the following criteria:

* Surgically sterile
* Willing to abstain from sexual intercourse or use a reliable form of contraception (e.g. condom), if having sex with a pregnant or non-pregnant woman of childbearing potential, from screening until 3 months after the final dose of IMP.
* Surgically sterilised or post-menopausal female partner or same-sex relationship.

Exclusion Criteria:

1. Liver disease other than chronic hepatitis B (a diagnosis of steatosis is permitted providing inclusion criterion 6 is met).
2. Evidence of Liver cirrhosis on Fibroscan screening (Liver cirrhosis is defined as a Fibroscan measurement of >11.5 KPa), or previous history or evidence of cirrhosis on radiological imaging, Fibroscan or liver biopsy.
3. Positive serology for HIV-1 or HIV-2 or HCV or HDV antibodies.
4. Immunodeficient or autoimmune conditions due to disease or medication e.g. systemic steroids within previous 12 weeks. (Topical or inhaled steroids are permissible).
5. Clinically relevant co-morbidity, e.g. autoimmune disease.
6. Clinically relevant anaemia or leukopenia in the opinion of the investigator.
7. Cancer or treatment for cancer within 3 years prior to screening excluding basal cell carcinoma of the skin, which is allowed.
8. Known or suspected intolerance or hypersensitivity to the IMP or closely related compounds or any of the stated ingredients.
9. Receipt of any IMP within 90 days prior to screening or currently receiving IMP or intent to receive IMP.
10. Current substance or alcohol abuse that in the opinion of the Investigator would interfere with compliance or with interpretation of study results.
11. Any condition that in the opinion of the Investigator might interfere with study objectives.
12. Pregnant or breastfeeding.
13. Subjects should not have received, during the 6 month period prior to screening, any medications or other treatments that may adversely affect the immune system such as allergy injections, immunoglobulins, interferons, cytotoxic drugs or other drugs known to be frequently associated with significant major organ toxicity, or systemic corticosteroids (oral or injectable).

    Immunosuppressive treatment such as azathioprine or mercaptopurine is not permitted 6 months prior to screening.
14. Administration of live vaccines (such as live influenza vaccinations or live travel vaccinations) from 10 days prior to the screening visit until Day 85.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-10-13 (Actual); Study Completion 2018-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Thursz, MD, Principal Investigator — Imperial College London
Locations (21):
- South Korea (11):
  - Pusan National University Busan Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
- United Kingdom (10):
  - University Hospitals Birmingham NHS Foundation Trust, Queen Elizabeth Hospital, Birmingham
  - University Hospitals Bristol, Bristol
  - Barts and The London School of Medicine and Dentistry, Blizzard Institiue, London
  - King's College Hospital, London
  - Royal Free Hospital, London
  - St. George's Hospital and Medical School, London
  - Imperial College London - St Mary's Campus, London
  - Pennine Acute Hospitals, Manchester
  - Bradford Teaching Hospitals, Bradford Royal Infirmary, North Yorks
  - Queen's Medical Centre, Nottingham Hospital, Nottingham

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase 1, randomised, double-blind, placebo-controlled clinical trial to evaluate the safety, tolerability, and immunogenicity of Vaccine FP-02.2 in hepatitis B e-antigen (HBeAg)-negative patients chronically infected with HBV aged 18 to 65 years who had been receiving entecavir or tenofovir for ≥ 2 years
Pre-assignment Details: Subjects who met all inclusion and no exclusion criteria and provided written informed consent were enrolled within 28 days of Screening. Approximately 10 subjects were enrolled in each of 6 treatment groups in 3 sequential cohorts
Groups:
- Placebo: Placebo component administered by IM injection on Days 1, 29, and 57.
  Placebo: Placebo
Period: Overall Study
Arm/Group | Placebo | IC31® Adjuvant | FP-02.2 Low Dose | FP-02.2 Low Dose With IC31® Adjuvant | FP-02.2 High Dose | FP-02.2 High Dose With IC31® Adjuvant
Started | 10 | 10 | 10 | 10 | 10 | 11
Completed | 10 | 10 | 10 | 10 | 10 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo component administered by IM injection on Days 1, 29, and 57
  Placebo: Placebo
- Total: Total of all reporting groups
Arm/Group | Placebo | IC31® Adjuvant | FP-02.2 Low Dose | FP-02.2 Low Dose With IC31® Adjuvant | FP-02.2 High Dose | FP-02.2 High Dose With IC31® Adjuvant | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 11 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (9.62) | 50.9 (7.61) | 41.5 (6.75) | 50.0 (7.63) | 47.6 (6.96) | 48.9 (9.80) | 47.8 (8.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 1 | 0 | 3 | 3 | 13
  Male | 9 | 5 | 9 | 10 | 7 | 8 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 10 | 10 | 10 | 10 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  South Korea | 2 | 8 | 0 | 5 | 4 | 11 | 30
  United Kingdom | 8 | 2 | 10 | 5 | 6 | 0 | 31
Race [Count of Participants; unit: Participants]
  White | 1 | 0 | 1 | 1 | 0 | 0 | 3
  Black or African American | 1 | 0 | 3 | 1 | 1 | 0 | 6
  Asian | 3 | 9 | 5 | 7 | 7 | 11 | 42
  Other | 1 | 0 | 1 | 1 | 0 | 0 | 3
  Multiple | 4 | 1 | 0 | 0 | 2 | 0 | 7
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.1 (4.87) | 24.6 (3.91) | 26.6 (3.35) | 26.8 (3.48) | 26.6 (3.89) | 23.7 (1.99) | 25.9 (3.73)
Liver stiffness by Fibroscan [Mean (Standard Deviation); unit: kPa] — Normal liver stiffness values are between 2 and 6 kPa. Higher values indicate greater liver stiffness and more fibrosis. Significant fibrosis generally commences at approximately 8.5 kPa, cirrhosis generally commences at approximately 15 kPa, and cirrhosis with clinically significant portal hypertension generally commences at approximately 25 kPa.
  kPa | 5.8 (1.32) | 4.2 (1.24) | 4.9 (1.41) | 5.4 (1.34) | 6.1 (2.25) | 4.6 (1.06) | 5.2 (1.57)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs)
Description: Incidences of all TEAEs, IP related TEAEs, severe TEAEs, TEAEs leading to discontinuation of IP, and serious TEAEs,
Time Frame: Throughout the study to Day 85
Population: Safety population (all subjects who received IP)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | IC31® Adjuvant | FP-02.2 Low Dose | FP-02.2 Low Dose With IC31® Adjuvant | FP-02.2 High Dose | FP-02.2 High Dose With IC31® Adjuvant
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 11
Participants
  Any treatment emergent adverse event (TEAE) | 9 | 3 | 7 | 7 | 4 | 6
  Possibly treatment related TEAE | 3 | 1 | 5 | 5 | 1 | 1
  Severe TEAE | 0 | 0 | 0 | 1 | 0 | 0
  TEAE leading to IP discontinuation | 0 | 0 | 0 | 0 | 0 | 1
  Serious adverse event | 0 | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Number of Subjects With Local Injection Site Reactions
Description: Incidence of local injection site reactions occurring up to 7 days after each injection
Time Frame: Days 1 through 64
Population: Safety population (all subjects who received IP)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | IC31® Adjuvant | FP-02.2 Low Dose | FP-02.2 Low Dose With IC31® Adjuvant | FP-02.2 High Dose | FP-02.2 High Dose With IC31® Adjuvant
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 11
Participants
  Any injection site reaction | 2 | 1 | 6 | 6 | 5 | 5
  Burning sensation | 1 | 0 | 0 | 3 | 2 | 0
  Erythema/redness | 2 | 0 | 0 | 1 | 0 | 1
  Induration/hardening | 2 | 1 | 0 | 0 | 1 | 0
  Pain (without pressure) | 1 | 0 | 6 | 3 | 3 | 4
  Pain/tenderness (on pressure) | 2 | 0 | 5 | 4 | 5 | 1
  Swelling | 2 | 0 | 2 | 0 | 0 | 0
  Wheal(s) | 1 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Immunological Response
Description: IFN-gamma ELISpot assay specific for FP-02.2 peptides using cryopreserved PBMCs
Time Frame: Change from baseline to Day 85
Measure: Median (Full Range); unit: spot forming units/ 10^6 PBMC
Arm/Group | Placebo | IC31® Adjuvant | FP-02.2 Low Dose | FP-02.2 Low Dose With IC31® Adjuvant | FP-02.2 High Dose | FP-02.2 High Dose With IC31® Adjuvant
Number analyzed (Participants) | 9 | 6 | 5 | 7 | 9 | 5
spot forming units/ 10^6 PBMC | 166.7 [-6717 to 6692] | 1683.3 [67 to 17350] | 900 [-300 to 4158] | 5608.3 [0 to 17483] | 1433.3 [-7717 to 7833] | 4804.2 [293 to 10192]

ADVERSE EVENTS:
Time Frame: Throughout the study to day 85
Description: Treatment emergent adverse events
Groups:
- Placebo: Placebo component.
  Placebo: Placebo
- IC31® Adjuvant: IC31® Adjuvant alone.
  IC31® Adjuvant: IC31® Adjuvant
- FP-02.2 Low Dose: A low dose of the FP-02.2 vaccine.
  FP-02.2 Vaccine: Synthetic Peptide Hepatitis B Vaccine
- FP-02.2 Low Dose With IC31® Adjuvant: A low dose of the FP-02.2 vaccine with IC31® Adjuvant.
  FP-02.2 Vaccine: Synthetic Peptide Hepatitis B Vaccine
  IC31® Adjuvant: IC31® Adjuvant
- FP-02.2 High Dose: A high dose of the FP-02.2 vaccine.
  FP-02.2 Vaccine: Synthetic Peptide Hepatitis B Vaccine
- FP-02.2 High Dose With IC31® Adjuvant: A high dose of the FP-02.2 vaccine with IC31® Adjuvant.
  FP-02.2 Vaccine: Synthetic Peptide Hepatitis B Vaccine
  IC31® Adjuvant: IC31® Adjuvant
Arm/Group | Placebo | IC31® Adjuvant | FP-02.2 Low Dose | FP-02.2 Low Dose With IC31® Adjuvant | FP-02.2 High Dose | FP-02.2 High Dose With IC31® Adjuvant
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 1/11
Other Adverse Events (participants affected / at risk) | 9/10 | 3/10 | 7/10 | 7/10 | 4/10 | 5/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | IC31® Adjuvant (N=10) | FP-02.2 Low Dose (N=10) | FP-02.2 Low Dose With IC31® Adjuvant (N=10) | FP-02.2 High Dose (N=10) | FP-02.2 High Dose With IC31® Adjuvant (N=11)
Moderate infectious colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | IC31® Adjuvant (N=10) | FP-02.2 Low Dose (N=10) | FP-02.2 Low Dose With IC31® Adjuvant (N=10) | FP-02.2 High Dose (N=10) | FP-02.2 High Dose With IC31® Adjuvant (N=11)
Nervous System disorders (Nervous system disorders) | 1 (1) | 1 (1) | 3 (4) | 3 (5) | 2 (3) | 0 (0)
Infections and infestations (Infections and infestations) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 0 (0) | 3 (3)
General disorders and administration site conditions (General disorders) | 2 (4) | 1 (1) | 1 (3) | 2 (3) | 2 (5) | 2 (2)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 3 (4) | 2 (5) | 1 (3) | 0 (0)
Gastrointestinal disorders (Gastrointestinal disorders) | 6 (9) | 1 (2) | 1 (2) | 2 (2) | 1 (1) | 1 (1)
Investigations (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular disorders (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-08-11): https://cdn.clinicaltrials.gov/large-docs/97/NCT02496897/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-09): https://cdn.clinicaltrials.gov/large-docs/97/NCT02496897/SAP_001.pdf